CLINICAL TRIAL: NCT00602992
Title: Exploring the Role of 3T MRI in Gamma Knife Radiosurgery: A Pilot Study
Brief Title: Exploring the Role of 3T MRI in Gamma Knife Radiosurgery
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 06-0427-CE
Record Dates: First submitted 2007-09-19; First posted 2008-01-28 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Brain Metastases
Keywords: 3T MRI; Gamma Knife Radiosurgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Gamma Knife radiosurgery is a non-invasive technique for the delivery of a single, high dose of radiation to an intra-cranial target. MRI has an established and central role in the treatment planning process and assessment of response to intracranial radiosurgery. Increasing the field strength of MRI from 1.5T to 3T promises to improve the signal, and in turn the quality of images. However, the technology also introduces new limitations, and the role and safety of 3T MRI in the management of patients receiving radiosurgery has not yet been reported. In this pilot study, we will explore the spatial integrity, and incremental image-guidance utility of 3T MRI in patients receiving radiosurgery. The preliminary data acquired in this study will be instrumental to the judicious design and conduct of subsequent definitive clinical trials. Up to fifty patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to receive Gamma Knife radiosurgery will be eligible for enrollment on this study.

Exclusion Criteria:

* Age<18
* Contra-indications to 3T MRI, such as implanted metal devices or shrapnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have consented to Gamma Knife radiosurgery.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Menard, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada